CLINICAL TRIAL: NCT03860129
Title: Depth of Long Term ICU Sedation Under 0,5 MAC Isoflurane, Sevoflurane or Desflurane Using MIRUS, an Automated Delivery System for Volatile Anaesthetics
Brief Title: Different Volatile Anaesthetics and the Depth of Long Term ICU Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Martin Bellgardt, Prof. Dr. med. Thomas Weber, Director Anesthesiology department St. Josef-Hospitital, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RUB 4780-13-B
Record Dates: First submitted 2018-09-24; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Intensive Care Unit Syndrome
Keywords: inhalational Sedation
MeSH Terms: interventions — Isoflurane; Sevoflurane; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ISO (Other): Drug name: Isoflurane Dosage form: inhalational Dosage: ml/h Concentration: 0.5 MAC (0.5 Vol%)
  Interventions: Drug: Isoflurane
- SEVO (Other): Drug name: Sevoflurane Dosage form: inhalational Dosage: ml/h Concentration: 0.5 MAC (1.0 Vol%)
  Interventions: Drug: Sevoflurane
- DES (Other): Drug name: Desflurane Dosage form: inhalational Dosage: ml/h Concentration: 0.5 MAC (3.0 Vol%)
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Isoflurane — Group A: Isoflurane (0.5 MAC)
  Other Names: Forene
  Arms: ISO
Drug: Sevoflurane — Group B: Sevoflurane (0.5 MAC)
  Other Names: Sevorane
  Arms: SEVO
Drug: Desflurane — Group C: Desflurane (0.5 MAC)
  Other Names: Suprane
  Arms: DES

SUMMARY:
The MIRUS system (TIM, Andernach, Germany) as well as the AnaConDa uses a reflector to conserve volatile anaesthetics (VA). Both systems can be paired with ICU ventilators, but MIRUS features an automated control of end-tidal VA concentrations (etVA). We compare depth of 0.5 MAC inhalational long-term sedation with Isoflurane (ISO), Sevoflurane (SEVO) or Desflurane (DES).

DETAILED DESCRIPTION:
The study was approved by the appropriate Institutional Review Board. Thirty ASA II-IV patients, undergoing elective or emergency surgery under general anaesthesia were included and randomized into three equal groups: ISO, SEVO or DES. We used MIRUS, a gas delivery system with a VA reflector, just like AnaConDa, that can be paired with common ICU ventilators. Additionally, MIRUS features the unique ability to maintain the end-tidal concentration (etVA) in target by automatically adjusting the delivery rate. Every 8 hours, the RASS was assessed by the nurse. The log of the EEG-Narcotrend Index (NI) was also included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Signing of the informed consent document (patient or relatives).
* Patient age 18 years or older.
* ASA I-III

Exclusion Criteria:

* ASA IV patients
* Epidural or spinal analgesia
* Allergy or known hypersensitivity to any of the study drugs
* Patients with known or suspected genetic susceptibility to malignant hyperthermia
* Previous participation in this trial
* Participation in another clinical trial within 4 weeks prior to selection.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12-10 (Actual); Primary Completion 2017-05-05 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
usage of volatile anesthetics at 0.5 MAC during ICU Sedation | up to one week
  Comparison between Isofluarne, Sevoflurane and Desflurane

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Weber, PhD, Principal Investigator — Ruhr University of Bochum, Germany

REFERENCES:
- [Background] Bomberg H, Glas M, Groesdonk VH, Bellgardt M, Schwarz J, Volk T, Meiser A. A novel device for target controlled administration and reflection of desflurane--the Mirus. Anaesthesia. 2014 Nov;69(11):1241-50. doi: 10.1111/anae.12798. Epub 2014 Jul 9. PMID 25040673
- [Background] Romagnoli S, Chelazzi C, Villa G, Zagli G, Benvenuti F, Mancinelli P, Arcangeli G, Dugheri S, Bonari A, Tofani L, Belardinelli A, De Gaudio AR. The New MIRUS System for Short-Term Sedation in Postsurgical ICU Patients. Crit Care Med. 2017 Sep;45(9):e925-e931. doi: 10.1097/CCM.0000000000002465. PMID 28441236
- [Background] Bellgardt M, Drees D, Vinnikov V, Procopiuc L, Meiser A, Bomberg H, Gude P, Vogelsang H, Weber TP, Herzog-Niescery J. Use of the MIRUS system for general anaesthesia during surgery: a comparison of isoflurane, sevoflurane and desflurane. J Clin Monit Comput. 2018 Aug;32(4):623-627. doi: 10.1007/s10877-018-0138-z. Epub 2018 Apr 9. PMID 29633099
- [Derived] Georgevici AI, Kyprianou T, Herzog-Niescery J, Procopiuc L, Loganathan S, Weber TP, Bellgardt M. Negative drift of sedation depth in critically ill patients receiving constant minimum alveolar concentration of isoflurane, sevoflurane, or desflurane: a randomized controlled trial. Crit Care. 2021 Apr 13;25(1):141. doi: 10.1186/s13054-021-03556-y. PMID 33849618
- [Derived] Bellgardt M, Georgevici AI, Klutzny M, Drees D, Meiser A, Gude P, Vogelsang H, Weber TP, Herzog-Niescery J. Use of MIRUS for MAC-driven application of isoflurane, sevoflurane, and desflurane in postoperative ICU patients: a randomized controlled trial. Ann Intensive Care. 2019 Oct 16;9(1):118. doi: 10.1186/s13613-019-0594-8. PMID 31620921